CLINICAL TRIAL: NCT01245699
Title: MIHS Emergency Department CPR Quality Improvement Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valleywise Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-037
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest, CPR, quality improvement
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Chest Compression before and after RealCPRHelp
Oversight: Data Monitoring Committee: No

ARMS (2):
- Before RTAVF and post-event debriefing (No Intervention): Before scenario-based training, real-time audiovisual CPR feedback, and post-event debriefing
- After RTAVF and post-event debriefing (Active Comparator): After scenario-based training, real-time audiovisual CPR feedback, and post-event debriefing
  Interventions: Behavioral: scenario-based training, real-time audiovisual CPR feedback, and post-event debriefing

INTERVENTIONS:
Behavioral: scenario-based training, real-time audiovisual CPR feedback, and post-event debriefing — scenario-based training for CPR, real-time audiovisual CPR feedback using R Series monitor-defibrillator during treatment, and post-event debriefing
  Arms: After RTAVF and post-event debriefing

SUMMARY:
The investigators will quantify the quality of chest compressions provided in the Emergency Department and determine whether the quality of chest compressions is related to patient outcome. The quality of chest compressions and patient outcomes will be assessed both before and after the introduction of audiovisual feedback in real time.

DETAILED DESCRIPTION:
The Emergency Department will be using E-series unit manufactured by ZOLL Medical Group (Chelmsford, MA). These units are equipped with an accelerometer-based system that allows for measurement of chest compression depth and rate. These units are also equipped with RealCPRHelp, and FDA-approved technology that provides real-time audiovisual feedback to providers on the quality of chest compressions.

In the first phase of the project, the ED providers will utilize the E-series units to treat all patients requiring chest compressions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older

Exclusion Criteria:

* less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2010-06-09 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2016-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bentley J Bobrow, MD, Principal Investigator — Valleywise Health
Locations (1):
- Maricopa Integrated Health System, Phoenix, Arizona, United States

REFERENCES:
- [Result] Bobrow BJ, Clark LL, Ewy GA, Chikani V, Sanders AB, Berg RA, Richman PB, Kern KB. Minimally interrupted cardiac resuscitation by emergency medical services for out-of-hospital cardiac arrest. JAMA. 2008 Mar 12;299(10):1158-65. doi: 10.1001/jama.299.10.1158. PMID 18334691

RESULTS

PARTICIPANT FLOW:
Groups:
- Before Training, RTAV CPR Feedback and Debriefing: Before scenario-based training, real-time audiovisual CPR feedback, and post-event debriefing
- After Training, RTAV CPR Feedback, and Debriefing: After scenario-based training, real-time audiovisual CPR feedback, and post-event debriefing.
Period: Overall Study
Arm/Group | Before Training, RTAV CPR Feedback and Debriefing | After Training, RTAV CPR Feedback, and Debriefing
Started | 61 | 54
Completed | 52 | 49
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Before training
- Phase 2: After training.
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase 2 | Total
Number analyzed (Participants) | 52 | 49 | 101
Age, Customized [Mean (Full Range); unit: years]
  Mean Age of participants | 56 [47 to 72] | 60 [45 to 68] | 58 [45 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 8 | 27
  Male | 33 | 41 | 74

OUTCOME MEASURES:

1. Primary Outcome: CPR Quality-compression Depth
Description: Measurement of chest compression depth
Time Frame: during CPR
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Before Training: Before scenario-based training, real-time audiovisual CPR feedback, and post-event debriefing
- After Training.: After scenario-based training, real-time audiovisual CPR feedback, and post-event debriefing
Arm/Group | Before Training | After Training.
Number analyzed (Participants) | 52 | 49
mm | 46.7 [42.9 to 50.5] | 61.6 [58.7 to 64.4]

2. Primary Outcome: CPR Quality-percent of >51mm Compressions
Description: Percent of Chest Compressions greater than 51mm
Time Frame: during CPR
Measure: Median (95% Confidence Interval); unit: percentage of chest compressions >51mm
Arm/Group | Before Training | After Training
Number analyzed (Participants) | 52 | 49
percentage of chest compressions >51mm | 30.6 [18.3 to 42.9] | 87.4 [74.6 to 100.1]
Statistical Analysis 1: Comparison: Before Training vs After Training; Test type: Superiority; p < 0.001, Kruskal-Wallis

3. Primary Outcome: CPR Quality
Description: Chest Compression Release Velocity
Time Frame: during CPR
Measure: Mean (95% Confidence Interval); unit: mm/s
Arm/Group | Before Training | After Training
Number analyzed (Participants) | 52 | 49
mm/s | 314 [289 to 338] | 442 [422 to 462]
Statistical Analysis 1: Comparison: Before Training vs After Training; Test type: Superiority; p < 0.001, Kruskal-Wallis

4. Primary Outcome: CPR Quality-compression Fraction
Description: Chest Compression Fraction indicating the percentage of time in which chest compressions are done by rescuers during a cardiac arrest
Time Frame: During CPR
Measure: Median (95% Confidence Interval); unit: % of time chest compressions are done
Arm/Group | Before Training | After Training
Number analyzed (Participants) | 52 | 49
% of time chest compressions are done | 84.3 [80.8 to 87.7] | 88.4 [84.8 to 91.9]
Statistical Analysis 1: Comparison: Before Training vs After Training; Test type: Superiority; p = 0.1, Kruskal-Wallis

5. Primary Outcome: CPR Quality-Chest Compression Rate
Description: Mean Chest Compression Rate
Time Frame: During CPR
Measure: Mean (95% Confidence Interval); unit: CCs/min
Arm/Group | Before Training | After Training
Number analyzed (Participants) | 52 | 49
CCs/min | 125 [122 to 128] | 125 [122 to 127]
Statistical Analysis 1: Comparison: Before Training vs After Training; Test type: Superiority; p = 0.65, Kruskal-Wallis

6. Primary Outcome: CPR Quality- Pre-shock Pause
Description: Pre-shock pause: time from cessation of CPR to shock delivery
Time Frame: During CPR
Measure: Median (95% Confidence Interval); unit: sec
Arm/Group | Before Training | After Training
Number analyzed (Participants) | 52 | 49
sec | 9.7 [3.0 to 16.3] | 5.9 [0 to 13.9]

ADVERSE EVENTS:
Time Frame: During CPR administered for cardiac arrest a minimum of 15 minutes.
Arm/Group | Phase I | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49
Other Adverse Events (participants affected / at risk) | 0/52 | 0/49

LIMITATIONS AND CAVEATS:
11 study participants were eliminated because event data was not captured. A single-center, nonrandomized, non-blinded, study. The Hawthorne effect may have affected results. Variations in the level of training and proficiency of providers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes